CLINICAL TRIAL: NCT07255508
Title: Efficacy of Prostatic Arteries Embolization Using SQUIDPERI
Acronym: SQUID-PAE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Balt International (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP250088; 2025-A00926-43 (Other: ANSM (French National Agency for the Safety of Medicines and Health Products))
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: Benign Prostate Hypertrophy(BPH)
Keywords: Prostatic Artery Embolization; PAE; SQUIDPERI; Liquid Embolic Agent
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Prostatic Artery Embolization
  Interventions: Device: Liquid embolic agent

INTERVENTIONS:
Device: Liquid embolic agent — Prostatic Artery Embolization using a non-adhesive liquid embolic agent composed of an EVOH (ethylene-vinyl alcohol) copolymer dissolved in DMSO (dimethyl sulfoxide), with micronized tantalum powder suspended within it
  Other Names: Squid Peri

SUMMARY:
Prostatic Artery Embolization (PAE) is a recognized mini-invasive treatment of bothersome Lower Urinary Tract Symptoms (LUTS) related to Benign Prostatic Hyperplasia (BPH). Particle embolics are used almost exclusively for embolization, with wide variation in the type and size of particles showing similar performance and safety results. Even if its durability relies on multiple risk factors, LUTS recurrence-free survival probability decreases with years. It is demonstrated that recanalization of the native prostatic artery is found in 66% of patients experiencing LUTS recurrence. Artery recanalization after several months has been reported in embolization with microparticles. The investigators addressed this issue using the liquid embolic agent SQUIDPERI in a prospective cohort of patients undergoing rePAE and showed a good clinical success rate (76.7%) at 3 months. Since then, the investigators perform initial PAE using SQUIDPERI with good results.

The aim of SQUID-PAE study is to assess the efficacy of PAE using SQUIDPERI in an initial PAE setting in a multicenter prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patient scheduled for a PAE using SquidPERI as part of routine care
* Patient informed who signed the informed consent form
* French social security affiliation
* Good understanding of the French language

Exclusion Criteria:

* Patient unwilling or unlikely to comply with FU schedule
* Known severe allergy to iodine
* Known severe hepatic impairment
* Vulnerable patient populations (such as patient under guardianship, curatorship, deprived of liberty)
* Patient that already had a PAE
* Patient on AME (state medical aid)
* Participation in any interventional study involving human participants or being in the exclusion period at the end of a previous study involving human participants, if applicable

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nonvulnerable men suffering from LUTS related to BPH and eligible to PAE.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Clinical success at 3 months | Baseline and 3 months
  Rate of clinical success defined as an IPSS <18 at follow-up with a decrease from baseline > 25% AND a quality of life (QoL, last question of IPSS questionnaire) < 4 at follow-up with a decrease from baseline ≥ 1.

SECONDARY OUTCOMES:
Immediate technical success | Embolization procedure (baseline)
  Rate of immediate technical success. Immediate technical success is defined as an embolization of both lobes of the prostate using SQUID PERI.
Clinical success at 6 months | Baseline and 6 months
  Rate of clinical success defined as an IPSS <18 at follow-up with a decrease from baseline > 25% AND a quality of life (QoL, last question of IPSS questionnaire) < 4 at follow-up with a decrease from baseline ≥ 1.
Clinical success at 9 months | Baseline and 9 months
  Rate of clinical success defined as an IPSS <18 at follow-up with a decrease from baseline > 25% AND a quality of life (QoL, last question of IPSS questionnaire) < 4 at follow-up with a decrease from baseline ≥ 1.
Clinical success at 12 months | Baseline and 12 months
  Rate of clinical success defined as an IPSS <18 at follow-up with a decrease from baseline > 25% AND a quality of life (QoL, last question of IPSS questionnaire) < 4 at follow-up with a decrease from baseline ≥ 1.
IPSS at 3 months | Baseline and 3 months
  Change in IPSS score and subscores compared to baseline.
IPSS at 6 months | Baseline and 6 months
  Change in IPSS score and subscores compared to baseline.
IPSS at 9 months | Baseline and 9 months
  Change in IPSS score and subscores compared to baseline.
IPSS at 12 months | Baseline and 12 months
  Change in IPSS score and subscores compared to baseline.
QoL at 3 months | Baseline and 3 months
  Change in QoL score (last question of IPSS questionnaire) compared to baseline.
QoL at 6 months | Baseline and 6 months
  Change in QoL score (last question of IPSS questionnaire) compared to baseline.
QoL at 9 months | Baseline and 9 months
  Change in QoL score (last question of IPSS questionnaire) compared to baseline.
QoL at 12 months | Baseline and 12 months
  Change in QoL score (last question of IPSS questionnaire) compared to baseline.
IIEF-15 at 3 months | Baseline and 3 months
  Change in IIEF-15 score and subscores compared to baseline.
IIEF-15 at 6 months | Baseline and 6 months
  Change in IIEF-15 score and subscores compared to baseline.
IIEF-15 at 9 months | Baseline and 9 months
  Change in IIEF-15 score and subscores compared to baseline.
IIEF-15 at 12 months | Baseline and 12 months
  Change in IIEF-15 score and subscores compared to baseline.
Adverse events and serious adverse events | Up to 12 months
  Number of adverse events and serious adverse events.
Benign prostatic hyperplasia medication at baseline | Baseline
  Number of benign prostatic hyperplasia medication.
Benign prostatic hyperplasia medication at 3 months | 3 months
  Number of benign prostatic hyperplasia medication.
Re-intervention for benign prostatic hyperplasia at 12 months | Up to 12 months
  Rate of re-intervention for benign prostatic hyperplasia (surgery, prostatic artery embolization).

CONTACTS AND LOCATIONS:
Overall Officials: Marc SAPOVAL, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Hôpital Timone (Radiologie adultes et neuroradiologie), Marseille
  - Hôpital Arnaud de Villeneuve (Service Imagerie diagnostique et interventionnelle), Montpellier
  - Hôpital Européen Georges Pompidou - AP-HP (Radiologie Interventionnelle vasculaire et oncologique), Paris
  - Institut Cardiovasculaire de Strasbourg (ICS) - Clinique Rhena (Radiologie interventionnelle vasculaire et oncologique), Strasbourg

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision. Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation (GDPR).